CLINICAL TRIAL: NCT00675194
Title: A Prospective, Open, Comparative Multicentre Phase II Study for the Evaluation of Irinotecan and Capecitabine Versus Cisplatin and Capecitabine in Advanced Gastric Adenocarcinoma or Gastric-Oesophagal Junction
Brief Title: Efficacy of Irinotecan and Capecitabine Versus(vs) Cisplatin and Capecitabine in Patients With Esophago-Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC-ICE-2003
Record Dates: First submitted 2008-05-06; First posted 2008-05-08 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Gastric Cancer
Keywords: cisplatin; capecitabine; gastric; irinotecan; metastatic; chemotherapy
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis | interventions — Cisplatin; Irinotecan; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Cisplatin, Irinotecan, Capecitabine

SUMMARY:
The purpose of this study is to determine which Arm (capecitabine + irinotecan versus capecitabine + cisplatin) shows higher response rates in the treatment of advanced gastric-oesophagal cancer

Furthermore, comparison of progression-free survival, 1-year survival, Quality of Life and safety

DETAILED DESCRIPTION:
capecitabine + irinotecan versus capecitabine + cisplatin, as published by Kang et al. (ASCO 2006)

ELIGIBILITY:
Inclusion Criteria:

* gastric or gastric-oesophagal junction adenocarcinoma
* unidimensional measurable disease
* Karnofsky index >/=60%

Exclusion Criteria:

* prior chemo- or radiotherapy
* colorectal diseases
* brain metastases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2003-10; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
response rate

SECONDARY OUTCOMES:
safety
progression free survival
1 year survival
Quality of Life
Analysis of the dose and efficacy of Epoetin beta weekly in anaemic patients

CONTACTS AND LOCATIONS:
Overall Officials: Markus Moehler, MD, Principal Investigator — Johannes Gutenberg University Mainz
Locations (1):
- Johannes Gutenberg Universität , I. Medizinische Klinik und Polokilinik, Mainz, Germany